CLINICAL TRIAL: NCT06002854
Title: Comparison Of The Outcome Of Treatment of Microneedling With Autologous Platelet- Rich -Plasma Versus Microneedling With Topical Insulin In The Treatment Of Post Acne Atrophic Scars.
Brief Title: Comparison Of Outcome Of Microneedling With Autologous PRP Vs Microneedling With Topical Insulin In Treatment Of Post Acne Atrophic Scars.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Nazia Jabeen, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2022-GENL/252/JPMC
Record Dates: First submitted 2023-03-25; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: ATROPHIC ACNE SCARS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A Microneedling with PRP(platelete rich plasma) (Experimental)
  Interventions: Drug: PRP( platelet rich plasma) and Insulin human
- GROUP B Microneedling with topical INSULIN (Experimental)
  Interventions: Drug: PRP( platelet rich plasma) and Insulin human

INTERVENTIONS:
Drug: PRP( platelet rich plasma) and Insulin human — Microneedling with autologus PRP reduces inflammationin acne scars. Insulin human is a new topical drug which is used nowadays for acne scars as it is more effective in producing collagen formation as well as new blood vessel formation

SUMMARY:
Microneedling with topical INSULIN is a simple, effective tool for building body's new collagen layers and thus an alternative to all erosive techniques such as lasers, peels. The skin responds to fine punctures with the release of growth factors. 8 It is a safe procedure that can be performed in the office without complications, with a good cost-benefit because it is economically viable without any effect on patient's daily activities. 9

ELIGIBILITY:
Inclusion Criteria:

* postacne atrophic scars ≥ 2 on Goodman and Baron's acne scar-grading system
* Either gender.
* Age 20-50 years.

Exclusion Criteria:

* lactation and pregnancy
* skin cancers and infection
* photosensitivity like SLE ,XP
* use of RETINOIDS in last 6 months.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Topical Insulin R with microneedling versus Platelets rich plasma in atrophic acne scars | Efficacy will be assesed upto 4 months.
  Efficacy will be assessed by using Goodman and Baron Qualitative Scar Grading System

CONTACTS AND LOCATIONS:
Overall Officials: KHADIJA ASADULLAH, MBBS, Principal Investigator — JPMC; FAIZA INAM, FCPS, Principal Investigator — JPMC; PARISA SANAWAR, FCPS, Principal Investigator — JPMC
Locations (1):
- JPMC, Karachi, Sindh, Pakistan